CLINICAL TRIAL: NCT06663137
Title: An Open Label, Single Arm Study, to Evaluate the Safety and Efficacy of NDV01 KIT in Patients With High Grade Non Muscle Invasive Bladder Cancer (NMIBC)
Brief Title: Open Label Study to Evaluate the Safety and Efficacy of NDV01 KIT in High Grade NMIBC
Acronym: HGNMIBC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Relmada Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REL-NDV01-011
Record Dates: First submitted 2024-08-08; First posted 2024-10-29 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Non Muscle Invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Docetaxel; Gemcitabine

STUDY DESIGN:
Intervention Model Description: Open label, single arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NDV01 (Experimental): 1. Treatment phase: 6 biweekly instillations - six instillations on Days 1, 14, 28, 42, 56, and 70
  2. Maintenance phase: monthly administration - maintenance period of monthly treatments on Day 107, Day 140, Day 187, Day 220, Day 250, Day 287, Day 310, and Day 340
  A subject that fails to meet CR at PDE visit will undergo reinduction of 6 biweekly installations of NDV01, which will be followed by maintenance treatments per the protocol schedule.
  Interventions: Drug: NDV01 intravesical controlled release formulation of gemcitabine and docetaxel

INTERVENTIONS:
Drug: NDV01 intravesical controlled release formulation of gemcitabine and docetaxel — NDV01 is administered intravesically using a catheter.
  Other Names: Gemcitabine and docetaxel

SUMMARY:
This is a prospective, single-arm study evaluating the safety and efficacy of NDV01 KIT, a fixed-dose combination of gemcitabine HCl and docetaxel, administered via intravesical instillation in patients with high-grade Non-Muscle Invasive Bladder Cancer (NMIBC). NDV01 KIT includes 60 mL Carbopol Gel followed by 15 g NDV01 solution (gemcitabine HCl 1000 mg and docetaxel 40 mg), administered biweekly for six treatments, followed by monthly maintenance therapy for up to 12 months. The study includes a pharmacokinetic (PK) sub-study assessing systemic exposure to NDV01's active ingredients.

DETAILED DESCRIPTION:
Eligible patients who sign informed consent will receive intravesical treatment with NDV01 KIT, consisting of a sequential instillation of Carbopol Gel followed by NDV01 solution using a 14F urethral catheter. The treatment phase includes six instillations on Days 1, 14, 28, 42, 56, and 70. Primary Disease Evaluation (PDE) will be conducted on Day 100 (±3). Patients achieving a complete response may continue into a maintenance phase with monthly instillations through Month 12.

Maintenance period of monthly treatments on Day 107, Day 140, Day 187, Day 220, Day 250, Day 287, Day 310, and Day 340.

The Primary Disease Evaluation (PDE) will be performed on Study Day 100±3.

A subset of patients will participate in a PK sub-study involving up to 15 blood draws to assess systemic levels of gemcitabine and docetaxel during the first treatment cycle.

Primary Objectives:

Assess safety of NDV01 KIT through the study period. Evaluate the complete response (CR) rate in patients with high-grade NMIBC.

Secondary Objectives:

Assess the durability of CR. Evaluate event-free survival (defined as high-grade recurrence-free survival). Assess the durability of event-free survival. Determine incidence and time to cystectomy. Determine overall survival. Monitor response durability through long-term follow-up.

Exploratory Objective:

Evaluate pharmacokinetic parameters of NDV01 KIT in a subset of patients during the initial treatment phase.

A subject that fails to meet CR at PDE visit will undergo reinduction of 6 biweekly installations of NDV01, which will be followed by maintenance treatments per the protocol schedule.

ELIGIBILITY:
Subjects may participate in the study if they meet all the following criteria:

Inclusion criteria:

* Aged 18 - 80 years old
* Able to give informed consent
* Histologically confirmed diagnosis of high grade non-muscle invasive bladder cancer (NMIBC) - patients having high-grade disease at first evaluation after induction BCG alone (at least 5 of 6 doses) may qualify in the absence of disease progression.
* Participants must be ineligible for or have elected not to undergo radical cystectomy.
* Available for the whole duration of the study.
* Life expectancy >2 years, in the opinion of the investigator.
* Eastern Cooperative Oncology Group (ECOG) status 2 or less.
* Absence of concomitant upper tract urothelial carcinoma or urothelial carcinoma within the prostatic urethra. Freedom from upper tract disease (if clinically indicated) as indicated by no evidence of upper tract tumor by either intravenous pyelogram, retrograde pyelogram, computed tomography (CT) scan with or without urogram, or MRI with or without urogram performed within 6 months of enrolment.
* Patients with prostate cancer on active surveillance at low risk for progression, defined as Prostate-Specific Antigen (PSA) < 10 ng/dL, Gleason score 6 and clinical stage tumor-1 (cT1) are permitted to be in the study at the discretion of the investigator (see exclusion criterion 10).
* Female patients of childbearing potential must use maximally effective birth control during the period of therapy, must be willing to use contraception for 1 month following the last study drug infusion and must have a negative urine or serum pregnancy test upon entry into this study. Otherwise, female patients must be postmenopausal (no menstrual period for a minimum of 12 months) or surgically sterile. 'Maximally effective birth control' means that the patient, if sexually active, should be using a combination of two methods of birth control that are approved and recognized to be effective by Regulatory Agencies.

Exclusion criteria:

* Current or previous evidence of muscle invasive (muscularis propria) or metastatic disease presented. Examples that increase the risk of metastatic disease are (but not limited to):
* Presence of lymphovascular invasion and/micropapillary disease as shown in the histology of the biopsy sample.
* Patients with T1 disease accompanied by the presence of hydronephrosis secondary to the primary tumor - Unless scheduled for treatment like nephrostomy or JJ stent insertion..
* Current systemic therapy for bladder cancer.
* Symptomatic urinary tract infection or bacterial cystitis (once satisfactorily treated, patients can enter the study).
* Clinically significant and unexplained elevated liver or renal function tests.
* Women who are pregnant or lactating or refuse to commit to using contraception anytime during the study.
* Any other significant disease or other clinical findings which in the investigator's opinion would prevent study entry.
* History of malignancy of other organ system within past 5 years, except treated basal cell carcinoma or squamous cell carcinoma of the skin and ≤ pathological tumor-2 (pT2) upper tract urothelial carcinoma at least 24 months after nephroureterectomy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Complete Response (CR) in High-Grade NMIBC | 48 weeks
  Complete response is defined by at least one of the following criteria:
  Negative cystoscopy and negative or atypical urine cytology; and/or Positive cystoscopy with biopsy-confirmed benign or low-grade NMIBC, along with negative urine cytology.
Frequency and severity of Adverse Events (AEs), including Serious Adverse Events (SAEs) and Treatment-emergent AEs (TEAEs) occurring at any time during the study Serious Adverse Events (SAEs) Treatment-Emergent Adverse Events (TEAEs) | 48 weeks
  Any new Change from Baseline to End of Study (EOS) in investigators assessment

SECONDARY OUTCOMES:
Durability of Complete Response (CR) in High-Grade NMIBC | 48 weeks
  Evaluate how long patients maintain CR over time.
Number of Patients with CR Among Those with Carcinoma In Situ (CIS) | 48 weeks
  Includes those with or without co-existing high-grade Ta or T1 papillary disease.
Incidence of Event-Free Survival (EFS) at 12 Months | 48 weeks
  Event-free survival is defined as survival without recurrence of high-grade disease.
Durability of event-free survival in patients with high-grade Ta or T1 papillary disease (without concomitant CIS), who have no recurrence of high-grade Ta or T1 papillary disease | 48 weeks
  Tumor recurrence

OTHER OUTCOMES:
Pharmacokinetic parameters of NDV01 KIT will be evaluated | 20 weeks
  PK measurement expressed as maximum plasma concentration for NDV01 and PK measurement expressed as half-life and area under curve for NDV01 Pharmacokinetic (PK).

CONTACTS AND LOCATIONS:
Overall Officials: Boris Chertin, Principal Investigator — Head of Urology Dep Share Tzedek Medical Center
Locations (1):
- Relmada Site, Raanana, Israel

IPD SHARING:
Plan to Share IPD: No
Not yet